CLINICAL TRIAL: NCT06962579
Title: The Effect of Personalized Exercise Interventions for the Prevention of Chemotherapy-induced Peripheral Neuropathy
Acronym: CIPN-EX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: University Hospital, Antwerp (Other); Universitaire Ziekenhuizen KU Leuven (Other); Kom Op Tegen Kanker (Other)
Responsible Party: Principal Investigator, Lore Dams, Dr., Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6776; Edge 3857 (Other: UZ Antwerpen (UZA)); S69491 (Other: UZ/KU Leuven)
Record Dates: First submitted 2025-04-13; First posted 2025-05-08 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy (CIPN)
Keywords: chemotherapy induced peripheral neuropathy; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): Participants receive a 12-week individually tailored exercise program from the start of taxane- or platinum-based chemotherapy, in addition to the standard of care (advice on physical activity during cancer treatment)
  Interventions: Behavioral: Exercise intervention
- No formal exercise intervention (No Intervention): Standard of care (advice on physical activity during cancer treatment)

INTERVENTIONS:
Behavioral: Exercise intervention — * 30-minute face-to-face session with physiotherapist outlining the state of the science on the importance and benefits of physical activity during and after cancer treatment and advising patients to engage in regular physical activity according to the general guidelines
  * 12-week individually tailored exercise program
    * Home-based aerobic exercise, 3 times per week at moderate intensity
    * Supervised resistance and sensorimotor exercises, 2 times per week
  Arms: Exercise intervention

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a debilitating and common side effect of neurotoxic cancer treatment. The most frequent symptoms include sensory disturbances and weakness in the hands and/or feet. CIPN can interfere with both daily activities and cancer treatment itself. Although there is proof of concept for physical activity as a preventive measure for CIPN, physical activity is currently not included in the international evidence-based guideline for the prevention of CIPN due to the need of larger sample-sized definitive studies. The aim of this project is, on the one hand, to investigate the preventive effect of an exercise program based on international physical activity guidelines on CIPN symptoms in patients with breast or colorectal cancer undergoing taxane- or platinum-based chemotherapy. On the other hand, the study will also explore how patients and healthcare professionals experience the implementation of physical activity during this phase of therapy. A prospective randomized controlled trial will be conducted, with CIPN symptoms as the primary outcome measure.

DETAILED DESCRIPTION:
The scientific goals of the project are:

1. The primary scientific objective of the study is to determine the effect of a patient-tailored exercise program based on exercise guidelines in oncology on sensory symptoms of CIPN (QLQ-CIPN20, sensory subscale) at short term (12 weeks) compared to usual care.
2. The secondary scientific objectives entail to examine if the exercise program has beneficial short (i.e., 12 weeks) and- or long term (i.e., 24 weeks) effects on symptoms of CIPN (QLQ-CIPN20, motor and autonomic subscale) and other biopsychosocial outcomes related to CIPN: (1) Signs of CIPN, (2) Physical functioning, (3) Psychosocial functioning, and (4) Relative dose intensity of chemotherapy.
3. The tertiary objective of this study is to perform a process evaluation. The aim of this process evaluation is to investigate the barriers and facilitators of the exercise program in patients receiving taxane- or platinum-based chemotherapy by examining adherence to the exercise program as well as how patients and healthcare providers perceive the implementation of the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* a primary diagnosis of breast, gynaecological or colon cancer, without distant metastasis
* been chemotherapy naïve
* been scheduled for at least 12 weeks of taxane- or platinum-based chemotherapy without other neurotoxic chemotherapy

Exclusion Criteria:

* life expectancy of less than six months according to the patient's oncologist or designee
* advanced stage of disease
* having a known current neuropathy
* having cognitive or physical limitations that contraindicate participation in a low- to moderate intensity home-based walking and progressive resistance program (determined by the patient's oncologist)
* not able to read and understand Dutch
* not able to provide informed consent
* not able to participate during the entire study period
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-induced peripheral neuropathy (CIPN) sensory symptom severity | at 12 weeks follow-up
  To evaluate the primary outcome sensory symptoms of CIPN, the Quality of Life Questionnaire-CIPN twenty-item scale will be used (QLQ-CIPN20 sensory subscale, score range from 9 to 36, higher scores indicating more sensory symptoms or problems).

SECONDARY OUTCOMES:
Chemotherapy-induced peripheral neuropathy (CIPN) sensory, motor and autonomic symptom severity | at 4, 8, 12 and 24 weeks follow-up
  To evaluate the sensory, motor and autonomic symptoms of CIPN, the Quality of Life Questionnaire-CIPN twenty-item scale will be used (QLQ-CIPN20). Each subscale score will be linearly transformed to a 0-100 scale with higher scores indicating greater symptom burden.
Relative dose intensity chemotherapy (%) | at 4, 8, 12 and 24 weeks follow-up
  Relative Dose Intensity (RDI) of chemotherapy, calculated as the ratio of delivered dose intensity to the planned dose intensity, expressed as a percentage.
Chemotherapy-induced peripheral neuropathy (CIPN) signs | at 12 and 24 weeks follow-up
  The Total Neuropathy Score clinical version (TNSc) is used to evaluate motor symptoms, pin sensation, vibration sensibility, tendon reflexes and strength in the hands and feet (score range 0-20, higher scores indicating greater severity of neuropathy).
Pain severity hands and feet | at 12 and 24 weeks follow-up
  Pain severity in the hands and feet will be evaluated with a Visual Analogue Scale (VAS). Four VAS scales will be completed: pain intensity at the present moment, mean pain intensity (global average pain intensity over the past week), maximum pain intensity (pain intensity at its maximum over the past week) and minimum pain intensity (pain intensity at its minimum over the past week).
General pain location and interference | at 12 and 24 weeks follow-up
  Pain location and pain interference will be evaluated with the Brief Pain Inventory (BPI), including a body diagram to identify painful body areas and a pain interference section measuring how pain impacts various aspects of daily life, including mood, sleep, work and social activities (score range 0-70, higher scores mean a worse outcome).
Physical functioning | at 12 and 24 weeks follow-up
  Evaluated with the PROMIS Short Form v2.0 Physical Function 8a questionnaire (scores expressed as T-scores with a mean of 50 (SD = 10) in the general population, higher scores mean a better outcome).
Self-reported physical activity | at 12 and 24 weeks follow-up
  Self-reported levels of physical activity are measured using the Godin-Shephard Leisure-Time Physical Activity Questionnaire.
Objective physical activity | at 12 and 24 weeks follow-up
  Minutes spent in different intensity zones (sedentary, light, moderate, vigorous) will be collected using a Fitbit device.
Fatigue | at 12 and 24 weeks follow-up
  Evaluated with the Multidimensional Fatigue Inventory (score range 20-100, higher scores mean a worse outcome).
Sleep disturbance | at 12 and 24 weeks follow-up
  Evaluated with the PROMIS Short Form v1.0 Sleep Disturbance 8a questionnaire (scores expressed as T-scores with a mean of 50 (SD = 10) in the general population, higher scores mean a worse outcome).
Depression | at 12 and 24 weeks follow-up
  Evaluated with the PROMIS Short Form v1.0 Depression 8a questionnaire (scores expressed as T-scores with a mean of 50 (SD = 10) in the general population, higher scores mean a worse outcome).
Anxiety | at 12 and 24 weeks follow-up
  Evaluated with the PROMIS Short Form v1.0 Anxiety 8a questionnaire (scores expressed as T-scores with a mean of 50 (SD = 10) in the general population, higher scores mean a worse outcome).
Social participation | at 12 and 24 weeks follow-up
  Evaluated with the PROMIS Short Form v2.0 Ability to participate in social roles and activities 8a questionnaire (scores expressed as T-scores with a mean of 50 (SD = 10) in the general population, higher scores mean a better outcome).
Support | at 12 and 24 weeks follow-up
  Evaluated with the PROMIS Short Form v2.0 Emotional support 4a, PROMIS Short Form v2.0 Instrumental support 4a and PROMIS Short Form v2.0 Informational support 4a questionnaires (scores expressed as T-scores with a mean of 50 (SD = 10) in the general population, higher scores mean a better outcome).
Cognitive function | at 12 and 24 weeks follow-up
  Evaluated with the Cognitive Failure Questionnaire (score range 0-100, higher scores mean a worse outcome).
Health-related quality of life | at 12 and 24 weeks follow-up
  Evaluated with the EuroQol-5Dimensions-5Levels (EQ-5D-5L) questionnaire, including the index score (based on the Belgian value set) and the EQ VAS (range 0-100), with higher scores indicating better health outcomes.

OTHER OUTCOMES:
Compliance - adherence to exercise intervention | From enrollment to the end of the intervention period at 12 weeks
  Evaluated with a self-composed questionnaire.
Beliefs about the efficacy of treatment | at 12 weeks follow-up
  Evaluated with the Patient Global Impression of Change questionnaire (score range 1-7, higher scores mean a worse outcome).
Safety of exercise intervention | From enrollment to the end of the intervention period at 12 weeks
  Evaluated with a self-composed questionnaire.
Patient experiences with exercise intervention | at 4, 8, 12 and 24 weeks follow-up
  Evaluated with a self-composed questionnaire.
Medication use | at 4, 8, 12 and 24 weeks follow-up
  Self-composed questionnaire.
Body Mass Index (BMI) | at 12 and 24 weeks follow-up
  BMI (kg/m²) will be calculated based on height (measured using a stadiometer) and weight (measured with the InBody 770 device).
Body composition - Extracellular water ratio | at 12 and 24 weeks follow-up
  The extracellular water to total body water ratio (ECW/TBW ratio) will be assessed using the InBody 770 bioimpedance analyzer.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - University Hospital Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Yes
The data are not openly available and are available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: On request
Access Criteria: On request